CLINICAL TRIAL: NCT02586402
Title: A Phase 2, Randomized, Active-controlled, Open-label, Multi-center Study of the Safety and Efficacy of Pegolsihematide for the Correction of Anemia in Patients With CRF Undergoing Dialysis and Previously Treated With ESAs
Brief Title: Safety & Efficacy of Pegolsihematide for Treatment of Anemia in Participants on Dialysis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-EPOP2c
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Renal Failure; Anemia; Dialysis
Keywords: ESAs CKD
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pegolsihematide (Experimental): Participants received Pegolsihematide by intravenous injection once every 4 weeks ; the dose was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 grams per deciliter (g/dL).
  Interventions: Drug: pegol-Sihematide
- Epoetin Alfa (Active Comparator): Epoetin Alfa administration 1 to 3 times per week. The dose was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: pegol-Sihematide
  Arms: Pegolsihematide
Drug: Epoetin Alfa
  Arms: Epoetin Alfa

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of multiple intravenous doses of pegol-Sihematide in participants with chronic kidney disease (CKD) who are on dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females≥18 and≤70, Weight ≥ 45 kilograms (kg)
2. Participants with chronic renal failure on dialysis for ≥ 3 months prior to randomization.
3. On ESAs treatment for ≥8 weeks prior to randomization with stable doses and the average doses ≤ 10000 IU/week
4. Hemoglobin values of ≥ 10.0 and≤ 12.0 g/dL at Screening
5. Patients with a transferrin saturation≥ 20% and a ferritin≥ 100 ng/mL. vitamin B12 and folic acid level above lower limit of normal.
6. Signed informed consent

Exclusion Criteria:

1. Pregnant or lactating females
2. Red blood cell transfusion within 3 months prior to randomization
3. Known intolerance to any erythropoiesis stimulating agent (ESA) or pegylated molecule or to all parenteral iron supplementation products
4. hemolytic syndromes or coagulation disorder
5. hematological disease (including but not limited to myelodysplastic syndrome, hematological malignancy, , hemoglobinopathy, pure red cell aplasia),
6. Chronic, uncontrolled, or symptomatic inflammatory disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, etc.);
7. C Reactive Protein (CRP) greater than 30 mg/L within the 4 weeks prior to randomization
8. Uncontrolled or symptomatic secondary hyperparathyroidism(iPTH>800pg/ml)
9. Poorly controlled hypertension within 4 weeks prior to randomization
10. Chronic congestive heart failure (New York Heart Association Class Ⅲ or IV)
11. significant symptom within 6 months prior to randomization (e.g. myocardial infarction, serious or precarious coronary artery disease,stroke, respiratory disease, autoimmune disease, neuropathy, phrenopathy, hepatopathy including Active hepatitis B, Active hepatitis C, A positive test for HIV antibody or ALT> 2 x upper limit of normal (ULN), AST> 2 x upper limit of normal (ULN))
12. tumor malignancy
13. Expected survival less than 12 months
14. A scheduled kidney transplant
15. Major surgery (may Massive bleeding) during the study
16. expected conception within 4 Weeks after the end of the Study Treatment
17. The subject has participated in other clinical trial within the 12 weeks prior to randomization
18. Have any other condition or prior therapy that, in the investigator's opinion, would make the subject unsuitable for the study, or unable or unwilling to comply with the study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Average reticulocytes and hemoglobin change from baseline | Baseline to Week 16

SECONDARY OUTCOMES:
Proportion of patients whose Hb within ±1.0 g/dL of baseline during Weeks 12 to 16 | week 12 to 16
Average RBC, hematokrit and reticulocytes change from baseline | Baseline to Week 16
Proportion of patients whose Hb levels were maintained within 10 to 12.0g/dL during Weeks 12 to 16 | week 12 to 16
Incidence of adverse events and serious adverse events | Baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Changli Mei, Study Chair — Changzheng Hospital
Locations (1):
- Changzheng Hospital, Shanghai, Shanghai Municipality, China